CLINICAL TRIAL: NCT02998580
Title: Conventional Bilateral rTMS vs. Bilateral Theta Burst Stimulation for Late-Life Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Daniel Blumberger, Principal Investigator, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 076-2016
Record Dates: First submitted 2016-12-16; First posted 2016-12-20 (Estimated); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Major Depression
Keywords: late-life depression; treatment resistance
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Convential Sequential Bilateral rTMS (Active Comparator): LFR followed by HFL.
  1 Hz stimulation of the right DLPFC for 600 pulses followed by 10 Hz stimulation of the left DLPFC for 3000 pulses (4 seconds on 26 seconds off for 75 trains). Treatment will occur 5 times per week for 4 to 6 weeks.
  Interventions: Device: LFR followed by HFL
- Bilateral Theta Burst Stimulation (Experimental): cTBS followed by iTBS.
  continuous theta burst stimulation (cTBS) of the right DLPFC for 600 pulses followed by intermittent theta burst stimulation (iTBS) of the left DLPFC for 600 pulses. Treatment will occur 5 times per week for 4 to 6 weeks.
  Interventions: Device: cTBS followed by iTBS

INTERVENTIONS:
Device: LFR followed by HFL — Magventure Cool B70 Coil with RX100 Stimulator
  Arms: Convential Sequential Bilateral rTMS
Device: cTBS followed by iTBS — Magventure Cool B70 Coil with RX100 Stimulator
  Arms: Bilateral Theta Burst Stimulation

SUMMARY:
This trial will compare conventional sequential bilateral rTMS to a bilateral theta burst stimulation protocol. The right and left dorsolateral prefrontal cortices will be the site of stimulation in both treatment conditions. The site of stimulation will be targeted using MRI co-registration. The study seeks to determine if the bilateral theta burst protocol has similar effectiveness to the conventional bilateral rTMS protocol in treating major depression.

ELIGIBILITY:
Inclusion Criteria:

* are an outpatient
* are ≥60 years old
* have a Mini-International Neuropsychiatric Interview (MINI 6.0)67 confirmed diagnosis of MDD, with a current MDE
* have failed to achieve a clinical response to an adequate dose of an antidepressant based on an Antidepressant Treatment History Form (ATHF) score of > 3 in the current episode or have failed to tolerate two separate trials of an antidepressant
* have a score > 17 on the MADRS
* have had no increase or initiation of any psychotropic medication in the 4 weeks prior to screening
* have normal electrolytes, hemoglobin and thyroid functioning based on pre-study blood work
* Pass the TMS adult safety screening (TASS) questionnaire
* Are able to have an MRI

Exclusion Criteria:

* have a history of substance dependence or abuse within the last 3 months
* have a concomitant major unstable medical illness determined by one of the study physicians
* have active suicidal intent
* have a lifetime MINI diagnosis of bipolar I or II disorder, or primary psychotic disorder
* have current psychotic symptoms
* have a diagnosis of obsessive compulsive disorder, post-traumatic stress disorder (current or within the last year), anxiety disorder (generalized anxiety disorder, social anxiety disorder, panic disorder), or dysthymia, assessed by a study investigator to be primary. One of these comorbidities will not be exclusionary if they are not deemed to be primary.
* have a diagnosis of any personality disorder, and assessed by a study investigator to be primary and causing greater impairment than MDD
* have presumed or probable dementia or clinical evidence of dementia as assessed by a Short Blessed Test score of greater than 10.
* did not respond to a course of ECT in the current depressive episode
* have received rTMS in the current episode, patients who have had rTMS in a previous episode would be eligible
* have a history of a primary seizure disorder or a seizure associated with an intracranial lesion.
* have an intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed
* have a implanted electronic device that is currently function such as a defibrillator
* currently take more than lorazepam 2 mg daily (or equivalent) or any dose of an anticonvulsant
* if participating in psychotherapy, must have been in stable treatment for at least 3 months prior to entry into the study, with no anticipation of change in the frequency of therapeutic sessions, or the therapeutic focus over the duration of the study
* non-correctable clinically significant sensory impairment (i.e., cannot hear well enough to cooperate with interview).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2020-04-24 (Actual); Study Completion 2020-04-24 (Actual)

PRIMARY OUTCOMES:
Change on the Montgomery Asberg Depression Rating Scale (MADRS) | After 4 or 6 weeks
  Change from baseline to week 4 or 6 endpoint

SECONDARY OUTCOMES:
Remission on the MADRS | After 4 or 6 weeks
  Score less than or equal to 10

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M. Blumberger, MD, Principal Investigator — CAMH
Locations (1):
- CAMH, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
The study protocol and statistical analysis plan will be made available. Individual patient data will be made available once all primary and secondary analyses have been conducted by the study team.
Supporting Information: Study Protocol, SAP
Time Frame: Individual patient data will be made available once all primary and secondary analyses have been conducted by the study team.

REFERENCES:
- [Derived] Adler E, Blumberger DM, Chen X, Lee HH, Nestor SM, Downar J, Mulsant B, Rajji TK, Noda Y, Daskalakis ZJ, Kaster TS. Trajectories of response to bilateral rTMS in late-life depression. Brain Stimul. 2025 Nov-Dec;18(6):2067-2074. doi: 10.1016/j.brs.2025.10.020. Epub 2025 Nov 1. PMID 41183728
- [Derived] Lee HH, Goke K, Wathra RA, Mulsant B, Trevizol AP, Downar J, McClintock SM, Nestor SM, Noda Y, Rajji TK, Daskalakis ZJ, Blumberger DM. Clinical effects and correlates of standard rTMS and theta burst stimulation (TBS) on suicidal ideation in late-life depression. Eur Psychiatry. 2025 Jun 27;68(1):e92. doi: 10.1192/j.eurpsy.2025.10049. PMID 40574540
- [Derived] Chen X, Blumberger DM, Yan CG, Downar J, Vila-Rodriguez F, Daskalakis ZJ, Kaster TS. Crosswalk between HRSD and MADRS outcomes for rTMS in patients with depression. BMJ Ment Health. 2025 Mar 28;28(1):e301451. doi: 10.1136/bmjment-2024-301451. PMID 40154967
- [Derived] Goke K, McClintock SM, Mah L, Rajji TK, Lee HH, Nestor SM, Downar J, Noda Y, Daskalakis ZJ, Mulsant BH, Blumberger DM. Cognitive Outcomes After Transcranial Magnetic Stimulation for the Treatment of Late-Life Depression: Resultats cognitifs apres la stimulation magnetique transcranienne pour le traitement de la depression chez les personnes agees. Can J Psychiatry. 2025 Jan 29:7067437251315515. doi: 10.1177/07067437251315515. Online ahead of print. PMID 39881587
- [Derived] Goke K, Trevizol AP, Ma C, Mah L, Rajji TK, Daskalakis ZJ, Downar J, McClintock SM, Nestor SM, Noda Y, Mulsant BH, Blumberger DM. Predictors of remission after repetitive transcranial magnetic stimulation for the treatment of late-life depression. Psychiatry Res. 2024 Apr;334:115822. doi: 10.1016/j.psychres.2024.115822. Epub 2024 Feb 29. PMID 38452496
- [Derived] Blumberger DM, Mulsant BH, Thorpe KE, McClintock SM, Konstantinou GN, Lee HH, Nestor SM, Noda Y, Rajji TK, Trevizol AP, Vila-Rodriguez F, Daskalakis ZJ, Downar J. Effectiveness of Standard Sequential Bilateral Repetitive Transcranial Magnetic Stimulation vs Bilateral Theta Burst Stimulation in Older Adults With Depression: The FOUR-D Randomized Noninferiority Clinical Trial. JAMA Psychiatry. 2022 Nov 1;79(11):1065-1073. doi: 10.1001/jamapsychiatry.2022.2862. PMID 36129719
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital, fully affiliated with the University of Toronto, and a PAHO/WHO Collab — http://www.camh.net/research